CLINICAL TRIAL: NCT00472758
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Dose-escalation, Multicenter Study to Evaluate the Safety and Tolerability of Single-Dose, Intravenously Administered MEDI-545, a Fully Human Anti-Interferon-Alpha Monoclonal Antibody, in Patients With Chronic Plaque Psoriasis
Brief Title: A Multicenter Study to Evaluate the Safety and Tolerability of Single-Dose for MEDI-545
Acronym: CP145
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP145
Record Dates: First submitted 2007-05-11; First posted 2007-05-14 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-11

CONDITIONS: Chronic Plaque Psoriasis
MeSH Terms: interventions — sifalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): MEDI 545
  Interventions: Biological: MEDI 545
- 2 (Placebo Comparator): Placebo IV
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: MEDI 545 — IV dosed at 1.0 mg/kg, 3.0,g/kg, 10.0mg/kg and 30.0mg/kg
  Arms: 1
Other: Placebo — IV Placebo dosed at 1.0 mg/kg, 3.0,g/kg, 10.0mg/kg and 30.0mg/kg
  Arms: 2

SUMMARY:
-To evaluate the safety and tolerability of a multiple doses of this drug in adult patients.

DETAILED DESCRIPTION:
-The primary objective of the study is to evaluate the safety and tolerability of escalating single IV doses of MEDI-545 in adult patients with chronic plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults, age 18 through 70 years of age at time of screening;
* Written informed consent obtained from the patient prior to receipt of any study medication or beginning study procedures;
* Documented clinical history of chronic plaque psoriasis;
* ≥ 3% body surface area (BSA) involvement in affected skin other than the face and scalp;
* Have at least two target plaques that are suitable for serial photographic assessments, one of which is of a size and location to allow serial biopsies;
* No significant changes in regular psoriasis treatment from at least 28 days from screening through the time of study drug administration;
* Sexually active women, unless surgically sterile or at least 1 year post-menopausal, must use an effective method of avoiding pregnancy (including oral, transdermal, or implanted contraceptives, intrauterine device, female condom with spermicide, diaphragm with spermicide, cervical cap, abstinence, use of a condom with spermicide by the sexual partner or sterile sexual partner) for 21 days prior to study drug administration, and must agree to continue using such precautions through Study Day 126. Cessation of birth control after this point should be discussed with a responsible physician. Sexually active men, unless surgically sterile, must likewise use an effective method of birth control (condom with spermicide) and must agree to continue using such precautions through Study Day 126;
* Willing to forego other forms of experimental treatment and study procedures during the study; and
* Ability to complete the study period, including follow-up period through Study Day 126.

Exclusion Criteria:

* Receipt of MEDI-545 in any previous clinical study;
* History of allergy or reaction to any component of the MEDI-545 formulation;
* Pustular, guttate, or erythrodermic psoriasis as the predominant disease type;
* Current use of potent topical corticosteroids, tacrolimus, or calcipotriol from 28 days prior to screening through study drug administration;
* Current use of phototherapy including tanning beds, Goeckerman or modified Goeckerman regimen, systemic corticosteroids, cyclosporin A, azathioprine, mycophenolate mofetil, methotrexate, or any other systemic treatment for psoriasis within 28 days prior to screening up through study drug administration;
* Current use of biologic agents such as alefacept or tumor necrosis factor-α inhibitors within 90 days prior to screening up through study drug administration;
* Any disease or illness, other than chronic plaque psoriasis, that may require the use of systemic corticosteroids during the study period;
* Acute illnesses or evidence of significant active infection, such as fever ≥ 38.0°C (≥ 100.5°F) from screening through study drug administration;
* Receipt of any investigational drug therapy or attenuated live vaccine therapy (other than vaccination against influenza) within 30 days or 5 half-life periods (whichever is longer) prior to study drug administration through the end of study;
* Pregnancy (sexually active women, unless surgically sterile or at least 1 year post-menopausal, must have a negative serum pregnancy test at screening and a negative urine pregnancy test prior to study drug administration on Study Day 0);
* Breastfeeding or lactating women;
* Evidence of infection with hepatitis B or C virus, or human immunodeficiency virus (HIV)-1 or -2, or active infection with hepatitis A, as determined by results of testing at screening;
* A history of severe infection with cytomegalovirus or viruses of the herpes family including Epstein-Barr virus requiring hospitalization, disseminated herpes, herpes encephalitis, or ophthalmic herpes;
* Herpes zoster within 3 months prior to screening;
* Current suppressive antiviral therapy for herpes or other viral infections;
* A history of cancer except basal cell carcinoma or in situ carcinoma of the cervix treated with apparent success with curative therapy ≥ 1 year prior to randomization;
* Elective surgery planned during the study period through end of study;
* Clinically significant abnormality, as determined by the investigator, on 12-lead electrocardiogram (ECG) or chest radiograph at screening;
* A history of coagulation disorders;
* History of primary immunodeficiency;
* History of stroke, or any cerebrovascular disease requiring current medication/treatment;
* In the opinion of the investigator, clinically significant active cardiac disease, including: unstable angina; myocardial infarction within 6 months; congestive heart failure; or arrhythmia requiring active therapy;
* Ongoing, clinically significant (in the opinion of the investigator) chronic infectious disease;
* History of active tuberculosis or positive tuberculosis (TB) test (defined as a reaction ≥ 10 mm in diameter) without a completed course of appropriate medical treatment;
* At the time of screening, any of the following: clinically significant abnormalities of hemoglobin, total white blood cell count, or platelet count; aspartate transaminase (AST) or alanine transaminase (ALT) > 1.5 times the upper limits of normal (ULN), serum creatinine, and prothrombin time (PT) or partial thromboplastin time (PTT) > ULN;
* Any other abnormal laboratory values in the screening panel that, in the opinion of the investigator, are clinically significant. Abnormal results on screening laboratory tests may be repeated once at the discretion of the site investigator(s) or qualified designee, prior to Study Day 0, to determine eligibility; or
* Evidence of any systemic disease or skin disease (other than chronic plaque psoriasis), any finding upon physical examination or history of any disease that, in the opinion of the investigator, designated health care provider, or medical monitor, may compromise the safety of the patient in the study or confound the analysis of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-02; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of MEDI-545 will be assessed through the collection of AEs and SAEs from study drug administration through Study Day 126. | Through day 26

SECONDARY OUTCOMES:
Secondary endpoints are the PK and IM of single-dose IV MEDI-545. | determination not stated

CONTACTS AND LOCATIONS:
Overall Officials: Barbara White, M.D., Study Director — MedImmune LLC
Locations (3):
- Canada (3):
  - Innovaderm Research, Laval, Inc., Laval-Quebec
  - Innovaderm Research, Inc., Montreal
  - Probity Medical Research, Waterloo- Ontario